CLINICAL TRIAL: NCT01416064
Title: Open-Label Extension Study to Evaluate the Safety of Molindone Hydrochloride Extended-Release Tablets as Adjunctive Therapy in Children With Impulsive Aggression Comorbid With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Open-Label, Extension Study to 810P202
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810P203
Record Dates: First submitted 2011-08-08; First posted 2011-08-12 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Impulsive Aggression Comorbid With ADHD in Children
MeSH Terms: interventions — Molindone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Molindone (Other): Extension study, all subjects will be given Molindone at different (established) dosage levels based on the patient's weight, response and investigator discretion.
  Interventions: Drug: Molindone

INTERVENTIONS:
Drug: Molindone — The populations will be comprised of male and female pediatric subjects from the 810P202 study. Subject will be converted to a total daily dose of 18 or 36mg of molindone (depending on weight), following enrollment into 810P203. The dosage level may be adjusted at the investigators discretion.

SUMMARY:
Open-label, extension study for subjects that completed 810P202 to examine long term safety and tolerability of repeated dosing of SPN-810M as an adjunctive therapy in children with Impulsive Aggression Comorbid with Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

1. Successful completion of the 810P202 study.
2. Continues to be medically healthy and with clinically normal laboratory profiles, vital signs, and electrocardiograms (ECGs).
3. Weight of at least 20kg.
4. Able and willing to swallow tablets whole and not chewed, cut or crushed.
5. Written informed consent/assent obtained from the subject's parent or legally-authorized representative (LAR), and written informed assent obtained from the subject if required.

Exclusion Criteria:

1. Body Mass Index (BMI) in 97th percentile or above.
2. Clinically significant change in health status that, in the opinion of the Investigator, would prevent the subject from participating in this study or successfully completing this study.
3. Pregnancy or refusal to practice contraception during the study (for female subjects of childbearing potential).
4. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study or complying with the study procedures.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Long Term Safety and tolerability of repeated oral dosing of 810M as an adjunctive therapy in children exhibiting impulsive aggression comorbid w/ ADHD | over 6 months
  Safety Assessments include: Adverse Events, clinical lab tests, vital signs, physical examinations, ECGs, Simpson-Angus Scale, Barnes Akathisia Scale, Abnormal Involuntary Movement Scale (AIMS) and Columbia Suicise Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Assess the efficacy of 810M | over 6 months
  Secondary efficacy endpoints: Retrospective-Modified Overt Aggression Scale (R-MOAS), Clinical Global Impression - Severity Scale (CGI-S), Clinical Global Impression - Improvement Scale (CGI-I), Swanson, Nolan and Pelman Rating Scale-Revised (SNAP-IV) ADHD scale scores

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Dothan, Alabama
  - Los Angeles, California
  - Santa Ana, California
  - Wildomar, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - North Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Libertyville, Illinois
  - Indianapolis, Indiana
  - Terre Haute, Indiana
  - Owensboro, Kentucky
  - Toms River, New Jersey
  - Stony Brook, New York
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Bellevue, Washington
  - Bothell, Washington